CLINICAL TRIAL: NCT04338815
Title: Exoskeleton Variability Optimization for Reducing Gait Variability for Patients With Peripheral Artery Disease
Brief Title: Exoskeleton Variability Optimization
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The second arm was not completed since the first arm was not successful based on the convergence criteria.
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0376-19-FB; P20GM109090 (NIH)
Record Dates: First submitted 2020-04-03; First posted 2020-04-08 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Arterial Disease
Keywords: Exoskeleton
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimal Assistance Pattern (Experimental): An optimization algorithm will change the assistance pattern on the hip exoskeleton during walking sessions and the optimal assistance pattern will be determined when gait variability is minimized.
  Interventions: Other: Exoskeleton Optimization
- Endurance Effectds (Experimental): Endurance of participants using ground reaction force (Bertec treadmill), walking speed (Bertec treadmill), indirect calorimetry (Cosmed), and motion capture (Vicon) will be determined.
  Interventions: Other: Endurance Evaluation

INTERVENTIONS:
Other: Exoskeleton Optimization — Participants will walk 10-minute trials while an optimization algorithm changes the assistance profile of the exoskeleton.
  Arms: Optimal Assistance Pattern
Other: Endurance Evaluation — Participants will walk 2 trials at a speed of 1 meter per second until the participant indicates claudication or a maximum duration of 6 minutes, which ever comes first.
  Arms: Endurance Effectds

SUMMARY:
Exoskeletons, wearable devices that assist with walking, can improve mobility in clinical populations. With exoskeletons, it is crucial to optimize the assistance profile. Recent studies describe algorithms (i.e., human-in-the-loop) to optimize the assistance profile with real-time metabolic measurements. The needed duration of current human-in-the-loop (HITL) algorithms range from 20 minutes to 1 hour which is longer than the average duration that most patients with peripheral artery disease (PAD) can walk. Because of this limited walking duration, it is often not possible for patients with PAD to reach steady-state metabolic cost, which makes these measurements are not useful for optimizing exoskeletons. In this study, investigators intend to develop and evaluate HITL optimization methods for exoskeletons and use the information to design and evaluate a portable hip exoskeleton. Shorter and more clinically feasible HITL optimization strategies based on experiments in healthy adults might allow utilizing these optimization strategies to become available for patient populations such as patients with PAD.

DETAILED DESCRIPTION:
Exoskeletons, wearable devices that assist with walking, can improve mobility in clinical populations. With exoskeletons, it is crucial to optimize the assistance profile. Recent studies describe algorithms (i.e., human-in-the-loop) to optimize the assistance profile with real-time metabolic measurements. The needed duration of current human-in-the-loop (HITL) algorithms range from 20 minutes to 1 hour which is longer than the average duration that most patients with peripheral artery disease (PAD) can walk. Because of this limited walking duration, it is often not possible for patients with PAD to reach steady-state metabolic cost, which makes these measurements are not useful for optimizing exoskeletons. Shorter and more clinically feasible HITL optimization strategies based on experiments in healthy adults might allow utilizing these optimization strategies to become available for patient populations such as patients with PAD.

This study will test different methods for optimizing exoskeletons. It will consist of an habituation session to the hip exoskeleton, an optimization session to find the optimal actuation settings using an algorithm that converges toward the optimum based on real-time measurements (human-in-the-loop algorithm) and a post-test at the end of optimization session to compare different conditions. The outcomes will be evaluated by surface electromyography, exoskeleton sensors, ground reaction force, walking speed, indirect calorimetry, and motion capture (Vicon).

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written consent
* Chronic claudication history
* Ankle-brachial index < 0.90 at rest
* Stable blood pressure, lipids, and diabetes for > 6 weeks
* Ability to walk on a treadmill for multiple five-minute spans
* Ability to fit in exoskeleton

  * Waist circumference 78 to 92 centimeters (31 to 36 inches)
  * Thigh circumference 48 to 60 centimeters (19 to 24 inches)
  * Minimal thigh length 28 centimeters (11 inches)

Exclusion Criteria:

* Resting pain or tissue loss due to peripheral artery disease (PAD, Fontaine stage III and IV)
* Foot ulceration
* Acute lower extremity event secondary to thromboembolic disease or acute trauma
* Walking capacity limited by diseases unrelated to PAD, such as:

  * Neurological disorders
  * Musculoskeletal disorders (arthritis, scoliosis, stroke, spinal injury, etc.)
  * History of ankle instability
  * Knee injury
  * Diagnosed joint laxity
  * Lower limb injury
  * Surgery within the past 12 months
  * Joint replacement
  * Pulmonary disease or breathing disorders
  * Cardiovascular disease
  * Vestibular disorder
* Acute injury or pain in lower extremity
* Current illness
* Inability to follow visual cues due to blindness
* Inability to follow auditory cues due to deafness
* Pregnant

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Malcolm, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No enrolled participants were tested in the endurance arm because the preceding optimal assistance arm was not successful based on the convergence criteria.
Groups:
- Optimal Assistance Pattern: An optimization algorithm will change the assistance pattern on the hip exoskeleton during walking sessions and the optimal assistance pattern will be determined when gait variability is minimized.
  Exoskeleton Optimization: Participants will walk 10-minute trials while an optimization algorithm changes the assistance profile of an exoskeleton.
- Effects on Endurance: The effects on endurance of participants using ground reaction force (Bertec treadmill), walking speed (Bertec treadmill), indirect calorimetry (Cosmed), and motion capture (Vicon) will be determined.
  Endurance Evaluation: Participants will walk 2 trials at a speed of 1 meter per second until the participant indicates claudication or a maximum duration of 6 minutes.
Period: Overall Study
Arm/Group | Optimal Assistance Pattern | Effects on Endurance
Started | 9 | 0
Completed | 0 | 0
Not Completed | 9 | 0

BASELINE CHARACTERISTICS:
Population: The effect on endurance arm was not analyzed since the preceding optimal assistance pattern aim was not successful based on the predefined convergence criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Optimal Assistance Pattern | Effects on Endurance | Total
Number analyzed (Participants) | 9 | 0 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 0 | 8
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 5 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 0 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Time to Convergence
Description: Convergence is determined when the estimated optimal exoskeleton settings vary less than 10%. The time to convergence is measured.
Time Frame: 10 minutes
Population: The time to convergence for the optimal assistance pattern could not be reported since the convergence criterion was not achieved. The effect on endurance arm was not analyzed since the preceding optimal assistance pattern aim was not successful based on the predefined convergence criteria.
Groups:
- Endurance Effectds: The effects on endurance of participants using ground reaction force (Bertec treadmill), walking speed (Bertec treadmill), indirect calorimetry (Cosmed), and motion capture (Vicon) will be determined.
  Endurance Evaluation: Participants will walk 2 trials at a speed of 1 meter per second until the participant indicates claudication or a maximum duration of 6 minutes.
Arm/Group | Optimal Assistance Pattern | Endurance Effectds
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Peak Extension Timing
Description: The time to peak extension moment of exoskeleton is measured by plotting the exoskeleton moment versus stride cycle percentage and finding the timing when the peak in the extension moment occurs expressed in percent of the stride cycle.
Time Frame: 20 seconds
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: % stride cycle
Arm/Group | Optimal Assistance Pattern | Effects on Endurance
Number analyzed (Participants) | 9 | 0
% stride cycle | 86 (8) |

3. Primary Outcome: Peak Flexion Timing
Description: The time to peak flexion moment of exoskeleton is measured by plotting the flexion moment versus stride cycle percentage and finding the timing when the peak in the flexion moment occurs expressed in percent of the stride cycle.
Time Frame: 20 seconds
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: % stride cycle
Arm/Group | Optimal Assistance Pattern | Effects on Endurance
Number analyzed (Participants) | 9 | 0
% stride cycle | 56 (2) |

4. Primary Outcome: Largest Lyapunov Exponent
Description: Largest Lyapunov exponent (the rate of separation of infinitesimally close trajectories) of lower limb kinematics is determined.
  Largest Lyapunov exponent is calculated using Wolf's algorithm. The theoretical range is from zero to plus infinity. Zero indicates an entirely stable periodic movement pattern. Higher values indicate more unstable and chaotic movement patterns. Lower values are considered better, and higher values are considered worse for gait stability.
Time Frame: 20 seconds
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: (Lyapunov exponent is unitless)
Arm/Group | Optimal Assistance Pattern | Effects on Endurance
Number analyzed (Participants) | 9 | 0
(Lyapunov exponent is unitless) | 6.6 (2.8) |

ADVERSE EVENTS:
Time Frame: 1.5 years
Description: The effect on endurance arm was not analyzed since the preceding optimal assistance pattern aim was not successful based on the predefined convergence criteria.
Arm/Group | Optimal Assistance Pattern | Effects on Endurance
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/0
Other Adverse Events (participants affected / at risk) | 0/9 | 0/0

LIMITATIONS AND CAVEATS:
The effect on endurance arm was not analyzed since the preceding optimal assistance pattern aim was not successful based on the predefined convergence criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT04338815/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT04338815/ICF_001.pdf